CLINICAL TRIAL: NCT02871687
Title: Effect of Statin Use on Aldosterone Secretion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jonathan S. Williams, MD, MMSc, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2016P000094
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Simvastatin; Pravastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo prepared by Investigational Drug Services at Brigham and Women's Hospital
  Interventions: Other: Placebo
- Simvastatin (Active Comparator): Subjects in the simvastatin arm will receive simvastatin 20 mg daily for 6 weeks before having their lipids checked. If their LDL-c decreases by less than 35% from screening, then the dose of simvastatin is increased to 40 mg daily for the following 6 weeks.
  Interventions: Drug: Simvastatin
- Pravastatin (Active Comparator): Subjects in the pravastatin arm will receive pravastatin 40 mg daily for 6 weeks before having their lipids checked. If their LDL-c decreases by less than 35% from screening, then the dose of pravastatin is increased to 80 mg daily for the following 6 weeks.
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 20 mg daily followed by potential increase to 40 mg simvastatin according to dose escalation procedure
  Other Names: Zocor
  Arms: Simvastatin
Drug: Pravastatin — Pravastatin 40 mg daily followed by potential increase to 80 mg pravastatin according to dose escalation procedure
  Other Names: Pravachol
  Arms: Pravastatin
Other: Placebo — Placebo prepared by Investigation Drug Services at Brigham and Women's Hospital
  Arms: Placebo

SUMMARY:
The purpose of this research protocol is to determine if the same effects are observed in vivo in humans through a randomized controlled study. Data regarding a novel mechanism of the widely used statin class of medications on the mineralocorticoid pathway would likely have significant clinical implications on the future management of hypertension and other cardiovascular disease given the known pleiotropy of aldosterone action.

DETAILED DESCRIPTION:
In order to provide additional evidence regarding the effect of statin therapy on aldosterone levels, the investigators propose the following randomized, double-blinded, placebo controlled protocol in relatively healthy volunteers. The investigators will evaluate aldosterone and cortisol production in response to an angiotensin II infusion under the following test conditions: 1) placebo, 2) simvastatin therapy (lipophilic statin), and 3) pravastatin therapy (hydrophilic statin). Measurements will be made to assess the effect of both acute (single dose) and chronic (6 and 12 weeks) therapy of the two statin medications.

ELIGIBILITY:
Inclusion Criteria:

* Blood pressure <140/90 mmHg and >90/50 mmHg
* Body mass index 19-40 kg/m2
* Normal screening laboratory values for:

  i. Serum sodium, potassium, glucose, liver enzymes ii. GFR (>60 mL/min/1.73m2) iii. A1c iv. TSH
* Normal ECG
* Negative urine HCG at screening for women who are able to become pregnant.

Exclusion Criteria:

* Any prior use of statin therapy
* History of coronary disease, diabetes, hypertension, stroke, kidney disease, thyroid disease, psychiatric illness, malignancy, preeclampsia, or illness requiring overnight hospitalization in the past 6 months
* Triglycerides > 500, LDL > 200
* Any prescription medication or herbal medication including oral contraceptive, excluding thyroid medications
* Unstable thyroid disease (determined by abnormal TSH)
* Pregnancy or current breastfeeding
* Alcohol intake >12 oz per week
* Tobacco or recreational drug use

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Serum aldosterone following angiotensin II infusion | 3 months

SECONDARY OUTCOMES:
24 hour urine aldosterone | Baseline
24 hour urine aldosterone | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Williams, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital- 221 Longwood Avenue, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baudrand R, Pojoga LH, Vaidya A, Garza AE, Vohringer PA, Jeunemaitre X, Hopkins PN, Yao TM, Williams J, Adler GK, Williams GH. Statin Use and Adrenal Aldosterone Production in Hypertensive and Diabetic Subjects. Circulation. 2015 Nov 10;132(19):1825-33. doi: 10.1161/CIRCULATIONAHA.115.016759. Epub 2015 Oct 2. PMID 26432671
- [Derived] Hornik ES, Altman-Merino AE, Koefoed AW, Meyer KM, Stone IB, Green JA, Williams GH, Adler GK, Williams JS. A clinical trial to evaluate the effect of statin use on lowering aldosterone levels. BMC Endocr Disord. 2020 Jul 14;20(1):105. doi: 10.1186/s12902-020-00587-4. PMID 32664962